CLINICAL TRIAL: NCT04451343
Title: The Life and Care of Patients With Colorectal Cancer Before Age 65 and Their Kindred
Acronym: MACHROAPIK
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MACHROAPICANCER
Record Dates: First submitted 2018-11-07; First posted 2020-06-30 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with a diagnosis of colorectal cancer before 65 years.
  Interventions: Other: biographical interviews
- Family: The spouse and /or children and /or parents of a patient 's diagnosis of colorectal cancer before 65 years.
  Interventions: Other: biographical interviews

INTERVENTIONS:
Other: biographical interviews — A sociologist trained in the sociology of cancer, to enable participants to talk about their experiences and clearly distinguish the experiences of each individual

SUMMARY:
In a context the respect of the autonomy of the patients is important, it is necessary to pay a sustained attention to the experiences and the lived experience as well of the patients suffering or in remission of cancer as of their family. It is therefore, for the family, to deepen the synthesis carried out by the Societal Cancer Observatory which is a societal observatory of cancer

ELIGIBILITY:
Inclusion Criteria:

Patients will be

* over 18 years old
* with a diagnosis of CRC before 65 years.
* able to give their non-opposition and to nominate at least 2 family members who would be willing to participate in the study

The spouse and / or children and / or parents will be eligible:

if they are at least 18 years old, if they can be considered a caregiver or are first-degree relatives of the index patient for whom a diagnosis of CRC has been made. .

Exclusion Criteria:

* Patients under 18 years of age or with a diagnosis of CRC after 65 years.
* Near a deceased patient or under 18 years old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surviving patients over the age of 18 and diagnosed with invasive CRC, infiltrating adenocarcinoma of the colon or rectum irrespective of the stage before 65 years old will be selected in the Poitou-Charentes cancer registry 2 to 5 years after announcement of the diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Assess the interaction between the care path (surgery, chemotherapy, radiotherapy) and the life course in patients before 65 years old with colorectal cancer | 2 hours
  semi-structured patients interview
Assess how the patients, their relatives and their family members, face the disease. | 1 hour
  semi-structured patients interview

CONTACTS AND LOCATIONS:
Locations (1):
- Registre du Cancer, Poitiers, France

IPD SHARING:
Plan to Share IPD: No